CLINICAL TRIAL: NCT04790734
Title: Efficacy and Safety of Remimazolam Besylate Versus Propofol for Sedation in Mechanically Ventilated ICU Patients: a Pilot Study
Brief Title: Efficacy and Safety of Remimazolam Besylate Versus Propofol for Sedation in Mechanically Ventilated ICU Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaobo Yang, MD, MD, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WUHICU202101
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Critical Illness
Keywords: Remimazolam besylate; Propofol; Intensive care unit; Mechanical ventilation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam (Experimental): Patients in the remimazolam group received remimazolam besylate at an initial infusion rate of 0.15 mg/kg/h and adjusted to maintain a RASS score of -3 to 0.
  Interventions: Drug: Sedation drugs
- Propofol (Active Comparator): Patients in the propofol group received propofol at an initial infusion rate of 2.0 mg/kg/h and adjusted to maintain a RASS score of -3 to 0.
  Interventions: Drug: Sedation drugs

INTERVENTIONS:
Drug: Sedation drugs — Different sedation drugs

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of remimazolam compared to propofol for sedation in mechanically ventilated ICU patients.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized, controlled pilot study using remimazolam and propofol for sedation in mechanically ventilated ICU patients. Subjects are randomized to remimazolam group and propofol group in a 1:1 ratio. Remifentanil is administered as the analgesic. Efficacy and safety profiles of remimazolam besylate are to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 75 years;
* Intubated and mechanically ventilated ≤96 hours before enrollment；
* Expected to require continuous invasive ventilation and sedation ≥24 hours;
* Requirement for light to moderate sedation (a RASS score of -3 to 0).

Exclusion Criteria:

* Body mass index (BMI) <18 or >30 kg/m2;
* Acute severe neurological disorder and any other condition interfering with RASS assessment;
* Systolic blood pressure less than 90 mm Hg after appropriate intravenous volume replacement and continuous infusions of 2 vasopressors;
* Heart rate less than 50 beats/min;
* Second- or third-degree heart block in the absence of a pacemaker;
* Unstable angina;
* Acute myocardial infarction;
* Left ventricular ejection fraction less than 30%;
* Contraindicate or allergic to study drugs;
* Moribund state;
* Acute hepatitis or serious hepatic dysfunction (Child-Pugh class C);
* Chronic kidney disease with glomerular filtration rate (GFR) < 60 ml/min/1.73m2;
* Alcohol abuse;
* Myasthenia gravis;
* Pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
The percentage of time in the target sedation range without rescue sedation | From the beginning of using study sedatives until being extubated, being discharged from our ICU, the study drug was stopped for 24 hours by physicians, or 7 days after enrollment, whichever came first
  The percentage of time in the target sedation range without rescue sedation

SECONDARY OUTCOMES:
Length of ICU stay | From start of study to 28 days
  Length of ICU stay
28-day mortality | From start of study to 28 days
  28-day mortality
7-day ventitlator free time | From start of study to 7 days
  7-day ventitlator free time

CONTACTS AND LOCATIONS:
Overall Officials: You Shang, Professor, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Critical Care Medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China

IPD SHARING:
Plan to Share IPD: No